CLINICAL TRIAL: NCT07100769
Title: Application of Real-time Ultrasound-guidance in Thoracic Epidural Catheter Placement on Patients Undergoing Major Abdominal Thoracic or Abdominal Surgeries
Brief Title: Application of Real-time Ultrasound Guidance in Thoracic Epidural Catheter Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/2025/HĐ-ĐHYD
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: First-attempt Success Rate of Real-time Ultrasound-guided Thoracic Epidural Catheter Placement
Keywords: Real-time ultrasound guided thoracic epidural catheter placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- real-time ultrasound guided thoracic epidural catheter placement (Experimental)
  Interventions: Procedure: Real-time ultrasound-guided thoracic epidural placement

INTERVENTIONS:
Procedure: Real-time ultrasound-guided thoracic epidural placement — Real-time ultrasound-guided thoracic epidural catheter placement is performed by an attending anesthesiologist using paramedian-cross view to approach thoracic epidural space.
  The patient is placed in the prone position with a pillow under the upper abdomen. The probe is placed to identify the rib, then moved medially to identify key anatomical structures: costotransverse joint, transverse process, lamina, superior articular process. The probe is rotated clockwise toward the midline to visualize the lamina and base of the spinal process.
  A 18G Tuohy needle is advanced under ultrasound guidance from inferior to superior aiming for the interspace between the lamina and base of the upper spinal process.
  After the tip of Tuohy needle approaches the interspace, the anesthesiologist will perform a loss-of-resistance test to identify the epidural space. Then a catheter will be inserted into epidural space.

SUMMARY:
The goal of this clinical trial is to assess the success rate of real-time ultrasound-guided thoracic epidural catheter placement at the first attempt in patients who will undergo thoracic or abdominal surgeries. The main aims are to:

Assess the success rate of first-attempt thoracic epidural catheter placement. Assess the procedure duration of real-time ultrasound-guided epidural catheter placement Participants will be managed according to the following protocol The patient will have real-time ultrasound guided catheter placement using paramedian-cross view performed by an attending anesthesiologist who is also an investigator After being secured, the thoracic epidural catheter is tested with 3ml lidocaine 2% At 30 minutes after the test dose, the level of sensory block is assessed by using an ice cube to test cold sensation on the skin according to dermatome Epidural analgesia is initiated by a 0.1ml/kg bolus and maintained by continuous infusion of solution 0.1% ropivacaine combined with 1mcg/ml fentanyl during the surgery At the end of the surgery, the patients will paracetamol 15miligram per kilogram and nefopam 20 milligrams, the patient will receive another epidural bolus dose of 0,1ml/kg ropivacaine 0.1% combined with fentanyl 1mcg/ml After the surgery, the patient will receive paracetamol 15miligram per kilogram every 8 hours, nefopam 20mg every eight hours, continuous epidural infusion at rate 4-8 ml per hour, patient-controlled analgesia morphine 1mg bolus, lockout 15 minutes, maximum 4mg per hour. Additional bolus dose of 4ml ropivacaine 0.1% will be administered every 30 min if VAS pain score at rest exceed 4. After two top-up bolus doses of 4ml ropivacaine 0.1% , if VAS pain score at rest still exceed 4, the patient will receive 2mg morphine every 15 minutes until VAS score less than 4 The patient will be monitored for vital signs, pain scores, the level of sensory block, opioids consumption, pain site, other adverse effect of opioids such as respiratory depression, sedation. The patient is also monitored for other signs and symptoms associated with nerve injuries or epidural hematoma such severe back pain, radicular pain, numbness, loss of sensation below the level of epidural catheter placement, paralysis or limb motor weakness.

DETAILED DESCRIPTION:
The consecutive sampling method is used in this clinical trial. Patients who meet inclusion criteria and consent to participate will be recruited Real-time ultrasound-guided epidural placement is performed by an attending anesthesiologists on participants using a paramedian-cross view to approach to the thoracic epidural space.

The process of real-time ultrasound-guided epidural catheter placement is described in detail in the following procedure.

Patient is placed in the prone position with continuous monitoring and oxygen supplementation via nasal cannula. A thin pillow is placed under the upper abdomen. After establishing an adequately sterilized field , the anesthesiologist places curvilinear probe on the 12th rib, then move cranially, until the rib below the target interlaminar space is reached. Then, probe is slid medially to identify anatomical structures: costotransverse joint, transverse process, lamina, superior articular process. Once consecutive laminas and superior articular processes are identified, the probe is the rotated clockwise toward the midline to visualize key ultrasound images from caudal to cranial positions: the lower transverse process, the lamina, the targeted interspace between the lower lamina and base of the upper spinal process. Then, 2ml of 1% lidocaine is administered to numb the anticipated skin puncture site. After that, 18G Tuohy needle is advanced under ultrasound guidance from inferior to superior aiming for the interspace between the lamina and base of the upper spinal process. Since the tip of Tuohy needle reaches the interspace between the lamina and base of the upper spinal process, the anesthesiologist performs a loss-of-resistance test using 0.9% saline to identify the thoracic epidural space. After achieving positive loss-of- resistance test, a catheter is advanced 4-5 cm into the epidural space. Finally, a test dose of 3 ml of 2% lidocaine is administered via the catheter.

At 30 minutes after the test dose, the level of sensory block is assessed by using an ice cube to test cold sensation on the skin. The evaluation will be conducted by an anesthesiologist or an anesthesia nurse. The cold sensation in the thoracic-abdominal dermatomes will be compared to the cold sensation in the shoulder or the ipsilateral arm and any reduction in cold perception in the tested dermatomes will be documented.

After having thoracic epidural catheter placement, the patient undergoes general anesthesia with routine monitoring. Intraoperative management is conducted by another attending anesthesiologist who doesn't participate in the study. After general anesthesia induction and patient positioning, the epidural catheter is activated with a bolus dose of 0.1 ml per kilogram solution of 0.1% ropivacaine + fentanyl 2mcg/ml. Vital signs are monitored every 5 minutes following epidural activation and for 15 minutes after surgical incision.

During the surgery, general anesthesia is maintained with sevoflurane or desflurane at MAC 1-1.2, along with continuous neuromuscular agent infusion to achieve TOF 0-1.The solution containing 0.1% ropivacaine and fentanyl 2mcg/ml at rate 4-8ml per hour is infused continuously via the epidural catheter. An additional intravenous bolus dose of fentanyl 1mcg/kg is administered if heart rate and blood pressure exceed 20% of baseline levels.

Before the completion of surgery, multimodal analgesia is initiated with intravenous paracetamol (15mg/kg) and nefopam (20mg). Additionally, a bolus dose of 0.1ml/kg of local anesthetic solution 0.1% ropivacaine combined with 2mcg/ml fentanyl is administered via the epidural catheter for postoperative pain control.

After surgery, patients will receive multimodal analgesia, including intravenous paracetamol 15 milligrams per kilogram and nefopam 20 milligrams every 8 hours. Epidural analgesia is maintained with a continuous infusion of 0.1% ropivacaine at a rate of 4-8 ml per hour, along with patient-controlled analgesia (PCA) morphine bolus dose of 1 milligram, with a 15-minute lockout interval and a maximum dose of 4 mg per hour.

Patients are monitored for vital signs, level of sensory blockade, pain scores using the Visual Analog Scale (VAS) at rest and during coughing, reported pain location, opioid consumption at specific time points 2, 8, 16, 24, and 48 hours postoperatively. If VAS pain scores at rest exceed 4, a top-up bolus of 4ml of 0.1% ropivacaine is administered via the epidural catheter. Vital signs, pain scores and the level of sensory block are monitored every 15 minutes following the rescue dose. A second 4ml 0.1% ropivacaine bolus can be administered 30 minutes after the first bolus. 30 minutes after the second, if the VAS score at rest still exceeds 4, a rescue 2mg morphine bolus every 15 minutes is administered until the VAS score is less than 4.

The epidural catheter is removed 48 hours after the surgery, provided there are no signs of severe back pain , neurological deficits, hypotension associated with epidural infusion, catheter dislodgement.

ELIGIBILITY:
Inclusion Criteria:

* Patients are scheduled for major thoracic or abdominal surgeries who have consented to thoracic epidural analgesia

Exclusion Criteria:

* Patients have contraindications for central neuraxial analgesia, allergic to medications used in the study, unable to cooperate due to cognitive impairment or behavioral limitations, spinal deformities or other spinal pathologies.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The first-attempt success rate of real-time ultrasound-guided thoracic epidural catheter placement | From skin puncture to successful thoracic epidural catheter placement
  The first-attempt success of thoracic epidural catheter placement is defined as success in achieving a positive loss-of- resistance test and placing the thoracic epidural catheter effortlessly after only one skin puncture
The procedure duration of real-time ultrasound-guided epidural catheter placement | From scanning to identify ultrasound image of the target structure to secure thoracic epidural catheter successfully
  The time duration from beginning to find ultrasound image of the target structure to successful thoracic epidural catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: PHAN TON NGOC VU, Phd, Principal Investigator — The University Medical Center Ho Chi Minh City
Locations (1):
- University Medical Center, Ho Chi Minh City, Ho Chi Minh City, Cho Lon, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Carvalho CC, Porto Genuino W, Vieira Morais MC, de Paiva Oliveira H, Rodrigues AI, El-Boghdadly K. Efficacy and safety of ultrasound-guided versus landmark-guided neuraxial puncture: a systematic review, network meta-analysis and trial sequential analysis of randomized clinical trials. Reg Anesth Pain Med. 2025 Sep 4;50(9):737-746. doi: 10.1136/rapm-2024-105547. PMID 38876801
- [Background] Kamimura Y, Yamamoto N, Shiroshita A, Miura T, Tsuji T, Someko H, Imai E, Kimura R, Sobue K. Comparative efficacy of ultrasound guidance or conventional anatomical landmarks for neuraxial puncture in adult patients: a systematic review and network meta-analysis. Br J Anaesth. 2024 May;132(5):1097-1111. doi: 10.1016/j.bja.2023.09.006. Epub 2023 Oct 6. PMID 37806932
- [Background] Deshmukh BY, Shetmahajan MG, Bakshi SG, Jain P. Predicting clinical entry point for thoracic epidural catheter insertion during paramedian approach: A prospective observational study. J Anaesthesiol Clin Pharmacol. 2024 Apr-Jun;40(2):248-252. doi: 10.4103/joacp.joacp_448_22. Epub 2024 Apr 26. PMID 38919420
- [Background] Hermanides J, Hollmann MW, Stevens MF, Lirk P. Failed epidural: causes and management. Br J Anaesth. 2012 Aug;109(2):144-54. doi: 10.1093/bja/aes214. Epub 2012 Jun 26. PMID 22735301
- [Background] Sivashanmugam T, Archana A, Nandhini P, Rani P. Real-time ultrasound-guided mid-thoracic epidural access using a novel paramedian cross (PX) view and drip infusion technique: a brief technical report. Reg Anesth Pain Med. 2024 Nov 4;49(11):840-844. doi: 10.1136/rapm-2023-105071. PMID 38388009